CLINICAL TRIAL: NCT06104722
Title: Comparison of the Effects of Copenhagen Adduction Exercise Performed at Different Loading Intensities on Hip Muscle Strength Development, Delayed Muscle Soreness, and Lower Extremity Physical Fitness Parameters
Brief Title: Comparison of the Effect of Copenhagen Adduction Exercises Performed at Different Load-intensity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ezgi Unuvar-Yuksel, principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: copenhagentkd2023
Record Dates: First submitted 2023-10-12; First posted 2023-10-27 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Groin Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high intensity copenhagen adduction exercise group (Experimental): Athletes in the high-intensity copenhagen adduction exercise group will perform classic copenhagen adduction exercise protocol.
  Interventions: Other: High-intensity Copenhagen adduction exercise
- low intensity copenhagen adduction exercise group (Experimental): Athletes in the low-intensity copenhagen adduction exercise group will perform a modified copenhagen adduction exercise protocol.
  Interventions: Other: Low-intensity Copenhagen adduction exercise

INTERVENTIONS:
Other: High-intensity Copenhagen adduction exercise — Copenhagen adduction exercise is an eccentric strengthening protocol of hip adductors and suitable for groin injury prevention and rehabilitation.
  Arms: high intensity copenhagen adduction exercise group
Other: Low-intensity Copenhagen adduction exercise — Copenhagen adduction exercise is an eccentric strengthening protocol of hip adductors and suitable for groin injury prevention and rehabilitation.
  Arms: low intensity copenhagen adduction exercise group

SUMMARY:
The aim of our study is to compare the effects of the Copenhagen adduction exercise, performed at different loading intensities, on hip muscle strength development, performance, flexibility, and delayed onset muscle soreness. The study will include active taekwondo athletes between the ages of 12-18. Athletes will be randomly divided into two groups: a low-intensity Copenhagen Adduction exercise group and a high-intensity Copenhagen Adduction exercise group. Athletes in both the low-intensity and high-intensity exercise groups will perform the exercise for 8 weeks in addition to their regular training program. At the beginning of the study and at the 4th, 8th, and 16th weeks, assessments will be conducted for hip abductor and adductor eccentric and isometric muscle strength, flexibility of the hip adductors, level of delayed muscle soreness, single-leg jump test, and timed lateral hop tests. The outcome of our study will determine how much improvement is achieved in hip muscle strength and lower extremity physical fitness parameters during and after the application of the Copenhagen adduction exercise at different loading intensities.

DETAILED DESCRIPTION:
The study is a single-blind randomized controlled trial including male and female adolescent taekwondo athletes (12-18 years). Evaluators will be blinded to which group are assessing.

Participants will be recruited from the local sports clubs. Club coaches will be asked to invite club players. Players interested in participating in the study will be asked to attend a meeting where the study will be explained to them. Those who were interested will then be assessed for inclusion and exclusion criteria.

Interventions:

Sports clubs are allocated to the high-intensity Copenhagen adductor exercise group (HCAE) or the low-intensity Copenhagen adduction exercise group (LCAE). Athletes in both the low-intensity and high-intensity exercise groups will perform the exercise for 8 weeks. Athletes in the HCAE group will perform the classic Copenhagen adduction exercise protocol and at LCAE group will perform the modified Copenhagen adduction exercise protocol.

Testing procedure:

The following tests will be performed before the exercise and 4th - 8th - 16th weeks after the beginning of the exercise.

The isometric and eccentric strength of the hip adductors and abductors Hip adduction flexibility Single-leg hop test Side hop test

A 10-point visual analog scale will be used to record the level of muscle soreness and rate of perceived exertion experienced after each training session.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 12-18
* Having a minimum of 3 years of experience as a taekwondo athlete
* Not having experienced any back, hip, or groin injuries in the last 12 months
* Participating in training sessions at least 3 days a week
* Being available to attend exercise training for 8 weeks

Exclusion Criteria:

* Having had a lower extremity orthopedic injury within the last 3 months
* Having an injury related to the hip and groin region
* Reporting a pain level of 4 or higher on the visual pain scale during the adductor squeeze test and palpation of the adductor muscles

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
hip muscle strength | beginning and 4th-8th-16th weeks after beginning
  isometric and eccentric hip adductor and abductor muscle strength will assess with a hand-held dynamometer.

SECONDARY OUTCOMES:
lower extremity performance | beginning and 4th-8th-16th weeks after beginning
  single leg hop test and side hop test
hip adduction flexibility | beginning and 4th-8th-16th weeks after beginning
  hip adduction range of motion will assess with a goniometer.
delayed onset muscle soreness | immediately after each exercise session, through 8 weeks
  delayed onset muscle soreness will assessed with visual analog scale.
rate of perceived exertion | immediately after each exercise session, through 8 weeks
  rate of perceived exertion will assessed with BORG CR10 scale(Borg Rating Of Perceived Exertion).

OTHER OUTCOMES:
exercise compliance | immediately after each exercise session, through 8 weeks
  participation status of all exercise session (%)

CONTACTS AND LOCATIONS:
Overall Officials: Hande Guney-Deniz, Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Altındag, Turkey (Türkiye)